CLINICAL TRIAL: NCT00776399
Title: Radiofrequency Ablation in Resectable Colorectal Lung Metastasis: A Phase-II Clinical Trial
Brief Title: Radiofrequency Ablation in Resectable Colorectal Lung Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mie University (Other)
Responsible Party: Principal Investigator, Koichiro Yamakado, instructor of Department of Interventional Radiology, Mie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-993 Mie-U-IRB
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Lung Metastasis; Colorectal Cancer
Keywords: Colorectal cancer; lung metastasis; radiofrequency ablation; metastasectomy; Lung metastasis from colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lung radiofrequency ablation (Experimental): A radiofrequency (RF) electrode is placed in the lung metastasis percutaneously. RF energy is applied to the tumor to induce coagulation necrosis.
  Interventions: Device: Lung radiofrequency ablation

INTERVENTIONS:
Device: Lung radiofrequency ablation — A radiofrequency (RF) electrode is placed in the lung metastasis percutaneously. RF energy is applied to the tumor to induce coagulation necrosis.
  Other Names: Cool-tip radiofrequency ablation system is used.

SUMMARY:
Lung metastasectomy is the only therapeutic option to provide a long-survival in patients with colorectal lung metastases. Recent studies have shown that radiofrequency (RF) ablation is a safe and useful therapeutic option for the treatment of unresectable lung metastases. In this phase-II trial, clinical utility of lung RF ablation will be evaluated in patients with resectable colorectal lung metastases.

DETAILED DESCRIPTION:
This will be a phase-II clinical trial.

Lung metastasectomy is the only therapeutic option to provide a long-survival in patients with colorectal lung metastases. Recent studies have shown that radiofrequency (RF) ablation is a safe and useful therapeutic option for the treatment of unresectable lung metastases. In this clinical trial, clinical utility of lung RF ablation will be evaluated.

Patients with resectable lung metastases will receive lung RF ablation.

All subjects will be followed for overall survival, safety, change in respiratory function, cancer-specific survival, and local tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Primary lesions (colorectal cancer) are resected.
* Lung metastases appear.
* No extrapulmonary metastases or after locoregional treatments.
* Lung metastasis is considered to be controllable either by metastasectomy or radiofrequency (RF) ablation.
* Five or less lung metastases measuring 3cm or smaller.
* PET study within 8 weeks before metastasectomy or RF ablation.
* White blood count of 3000/mm3 or more.
* Platelet count of 100,000/mm3 or more.
* Hemoglobin level of 8.0 g/dl.
* Serum creatinine level of 2.0 mg/dl or less.
* PaO2 of 70 mm Hg or more（Room air）or SpO2 of 93%.
* Serum bilirubin level of 2.0 mg/dl or less.
* Performance status of 0 or 1.
* Expected survival of 1 year or more.
* Age of 20 years or more.
* Informed consent from the patient.

Exclusion Criteria:

* Risk to injure lung vessels 5 mm or larger.
* Lung metastases adjacent to the heart, trachea, esophagus, and aorta.
* Association of uncontrollable malignancies.
* Lung hilar lymph node metastasis.
* One lung.
* Pulmonary hypertension.
* Coagulopathy.
* Impossible to stop using anticoagulants.
* Active infection or C-reactive protein of 3 or higher.
* Association of active inflammation.
* Fever (higher than 38 degrees celsius).
* Previous external-beam radiotherapy for the treated lung.
* Pregnant.
* Judgment to be an inappropriate candidate by a attending physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2017-12-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures:3-year survival | 3 years

SECONDARY OUTCOMES:
Secondary Outcome measures:safety, change in respiratory function, cancer-specific survival, and local tumor progression, Radiological studies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Haruyuki Takaki, MD, Study Director — Department of Radiology, Mie University School of Medicine
Locations (16):
- Japan (16):
  - Anjo kosei hospital, Anjo, Aichi-ken
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Hokkaido University, Sapporo, Hokkaido
  - Yamada red-cross hospital, Ise, Mie-ken
  - Matsusaka munipal hospital, Matsusaka, Mie-ken
  - Matsusaka central hospital, Matsusaka, Mie-ken
  - Suzuka Kaisei Hospital, Suzuka, Mie-ken
  - Suzuka central hospital, Suzuka, Mie-ken
  - Toyama hospital, Tsu, Mie-ken
  - Mie central medical center, Tsu, Mie-ken
  - Mie University, Tsu, Mie-ken
  - Mie prefectual medical center, Yokkaichi, Mie-ken
  - Okayama University, Kayama, Okayama-ken
  - Kumamoto University, Kumamoto
  - Kyoto Prefectual University of Kyoto, Kyoto
  - Okayama Saiseikai Hospital, Okayama

REFERENCES:
- [Background] Yamakado K, Hase S, Matsuoka T, Tanigawa N, Nakatsuka A, Takaki H, Takao M, Inoue Y, Kanazawa S, Inoue Y, Sawada S, Kusunoki M, Takeda K. Radiofrequency ablation for the treatment of unresectable lung metastases in patients with colorectal cancer: a multicenter study in Japan. J Vasc Interv Radiol. 2007 Mar;18(3):393-8. doi: 10.1016/j.jvir.2006.11.003. PMID 17377185
- [Derived] Hasegawa T, Takaki H, Kodama H, Yamanaka T, Nakatsuka A, Sato Y, Takao M, Katayama Y, Fukai I, Kato T, Tokui T, Tempaku H, Adachi K, Matsushima Y, Inaba Y, Yamakado K. Three-year Survival Rate after Radiofrequency Ablation for Surgically Resectable Colorectal Lung Metastases: A Prospective Multicenter Study. Radiology. 2020 Mar;294(3):686-695. doi: 10.1148/radiol.2020191272. Epub 2020 Jan 14. PMID 31934829